CLINICAL TRIAL: NCT00504439
Title: A Randomised, Double-blind, Placebo Controlled, Dose Ascending, Parallel Group Study to Evaluate the Safety, Tolerability, Steady State Pharmacokinetics and Pharmacodynamics of SB-656933-AAA Following Repeated Doses in Healthy Adult Subjects. The Pharmacokinetic Interaction Between Repeated Doses of SB-656933-AAA and Single Dose of Simvastatin Will Also be Assessed
Brief Title: A Study To Evaluate The Safety And Tolerability Of SB-656933-AAA Following Repeated Doses In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CR2100609
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD,; CD11b,; CXCR2,; safety,; repeat dose,; tolerability.; SB-656933,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — SB 656933; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive 20 milligrams (mg) of SB-656933-AAA once daily or matching placebo once daily for 14 days.
  Interventions: Drug: SB-656933-AAA; Drug: Matching placebo
- Cohort 2 (Experimental): Subjects will be administered 40 mg simvastatin on day 1 followed by a washout period of two days. From day 3, the subjects will receive 50 mg of SB-656933-AAA once daily or matching placebo once daily for 14 days. On day 17, subjects will be administered 40 mg simvastatin along with SB-656933-AAA to assess statin interaction.
  Interventions: Drug: SB-656933-AAA; Drug: Matching placebo; Drug: Simvastatin
- Cohort 3 (Experimental): Subjects will be administered 100 mg SB-656933-AAA/ day or matching placebo for 14 days. Dosing will initiate after cohort I and II have completed dosing.
  Interventions: Drug: SB-656933-AAA; Drug: Matching placebo

INTERVENTIONS:
Drug: SB-656933-AAA — The doses of SB-656933 (20 mg, 50 mg or 100 mg) will be provided as a combination of 10 mg and 50 mg tablets of SB-656933-AAA. The tablets will be administered orally.
  Other Names: SB-656933
Drug: Matching placebo — SB-656933-AAA matching placebo tablets will be administered orally.
Drug: Simvastatin — Simvastatin will be provided as a 40 mg tablet.
  Arms: Cohort 2

SUMMARY:
To assess safety of SB-656933 following repeat dosing for 14 days.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo controlled, dose ascending, parallel group study to evaluate the safety, tolerability, steady state pharmacokinetics and pharmacodynamics of SB-656933-AAA following repeated doses in healthy adult subjects. The pharmacokinetic interaction between repeated doses of SB-656933-AAA and single dose of simvastatin will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female, aged 18-65 years.
* Female must not be able to have children.
* Non-smoking for the last 6 months.

Exclusion Criteria:

* Any serious medical condition.
* Hepatitis B or C and/or HIV positive.
* Currently on HRT, or other medication except paracetamol.
* Body Mass Index >30.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-06-04 (Actual); Primary Completion 2007-09-06 (Actual); Study Completion 2007-09-06 (Actual)

PRIMARY OUTCOMES:
Assess safety of SB-656933 after repeat doses. | after repeat doses

SECONDARY OUTCOMES:
Investigate concentrations of SB-656933 in the body and how long it remains in the body over 14 days of repeat dosing. | 14 days of repeat dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study CR2100609 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CR2100609?search=study&search_terms=CR2100609#rs